CLINICAL TRIAL: NCT02525588
Title: Polyethylene Wear Study on the Triathlon Total Knee Prosthesis A Prospective Randomized Single Centre Roentgen Stereophotogrammetric Analysis (RSA) Study
Brief Title: Polyethylene Wear Study on the Triathlon Total Knee Prosthesis
Acronym: X3vsN2Vac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: K-S-039
Record Dates: First submitted 2015-06-11; First posted 2015-08-17 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional polyethylene inlay nitrogen/vacuum-packed (N2Vac) (Active Comparator): Conventional UHMWPE inlay in a Triathlon Condyle Stabilizing (CS) fixed bearing total knee prosthesis
  Interventions: Device: Triathlon CS fixed bearing total knee prosthesis
- Highly cross-linked polyethylene (X3) (Active Comparator): X3 highly cross-linked polyethylene inlay in a Triathlon CS fixed bearing total knee prosthesis
  Interventions: Device: Triathlon CS fixed bearing total knee prosthesis

INTERVENTIONS:
Device: Triathlon CS fixed bearing total knee prosthesis — The patient will receive either the N2Vac polyethylene inlay or the X3 polyethylene inlay for their CS total knee.

SUMMARY:
Comparison of conventional UHMWPE (ultra-high-molecular-weight polyethylene) with highly cross-linked polyethylene (X3) in a condylar stabilizing (CS) fixed bearing total knee prosthesis by means of RSA and clinical evaluation.

DETAILED DESCRIPTION:
The goal of this study is to compare conventional UHMWPE with X3 highly cross-linked polyethylene in a CS fixed bearing total knee prosthesis (Triathlon Knee System: Stryker, Warsaw, USA) by means of RSA and clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to understand the meaning of the study and is willing to sign the Ethic Commission approved, study specific Informed Patient Consent Form.
2. Patients with a pre-operative knee score of < 70.
3. Patients scheduled to undergo primary total knee replacement with any of the following indication.

   * Painful and disabled knee joint resulting from osteoarthritis.
   * One or more compartments are involved.
4. Need to obtain pain relief and improve function.
5. Ability and willingness to follow instructions, including control of weight and activity level, and to return for follow-up evaluations.
6. A good nutritional state of the patient.
7. Full skeletal maturity of the patient, patients who are at least 18 years of age.
8. Patients of either sex.

Exclusion Criteria:

1. The subject is morbidly obese, defined as Body Mass Index (BMI) of > 40.
2. Skeletal immaturity of the patient, patients who are less than 18 years of age.
3. Patient has a flexion contracture of 15° and more.
4. Patient has a varus/valgus contracture of 15° and more.
5. Patients with a pre-operative knee score of >70.
6. The subject has a history of total or unicompartmental reconstruction of the affected joint.
7. The subject will be operated bilaterally.
8. Patients who had a Total Hip Arthroplasty (THA) on contralateral and/or ipsilateral side within the last year that is considered to have an unsatisfactory outcome (Patients with contralateral and/or ipsilateral THA > 1 year ago with good outcome can be included in the study).
9. Patients who had a Total Knee Arthroplasty (TKA) on contralateral side within the last 6 months that is considered to have an unsatisfactory outcome. (Patients with contralateral TKA > 6 months ago with good outcome can be included in the study).
10. The subject has an active or suspected latent infection in or about the knee joint.
11. Osteomyelitis.
12. Sepsis.
13. Patients who will need lower limb joint replacement for another joint within one year.
14. The subject has a neuromuscular or neurosensory deficiency, which would limit the ability to assess the performance of the device.
15. The subject has a systemic or metabolic disorder leading to progressive bone deterioration.
16. The subject is immunologically suppressed or receiving steroids in excess of normal physiological requirements.
17. The subject's bone stock in compromised by disease or infection which cannot provide adequate support and/or fixation to the prosthesis.
18. The subject has had a knee fusion to the affected joint.
19. Female patients planning a pregnancy during the course of the study.
20. The patient is unable or unwilling to sign the Informed Consent specific to this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2019-03-28 (Actual); Study Completion 2019-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Kaptijn, MD, Principal Investigator — 't Langeland Ziekenhuis Zoetermeer
Locations (1):
- Department of Orthopaedics 't Langeland Ziekenhuis Zoetermeer, Zoetermeer, South Holland, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four patients were included into the study but not assigned to a group as prior to surgery two patients withdraw, one surgery was cancelled due to urinary tract infection and one patient met exclusion criteria BMI>40
Groups:
- N2Vac Polyethylene Inlay: Conventional UHMWPE inlay in a Triathlon CS fixed bearing total knee prosthesis
  Triathlon CS fixed bearing total knee prosthesis: The patient will receive either the N2Vac polyethylene inlay or the X3 polyethylene inlay for their CS total knee.
- X3 Highly Cross-linked Polyethylene: X3 highly cross-linked polyethylene inlay in a Triathlon CS fixed bearing total knee prosthesis
  Triathlon CS fixed bearing total knee prosthesis: The patient will receive either the N2Vac polyethylene inlay or the X3 polyethylene inlay for their CS total knee.
Period: Overall Study
Arm/Group | N2Vac Polyethylene Inlay | X3 Highly Cross-linked Polyethylene
Started | 48 | 48
Completed | 42 | 45
Not Completed | 6 | 3
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: Race or Ethnicity Baseline Measure is not captured in the Netherlands
Groups:
- Total: Total of all reporting groups
Arm/Group | N2Vac Polyethylene Inlay | X3 Highly Cross-linked Polyethylene | Total
Number analyzed (Participants) | 48 | 48 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.42 (10.24) | 64.31 (10.22) | 64.36 (10.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 32 | 63
  Male | 17 | 16 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 48 | 48 | 96
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.32 (4.18) | 29.61 (3.63) | 29.46 (3.90)
Indication [Count of Participants; unit: Participants]
  Osteoarthritis | 47 | 47 | 94
  Post Traumatic Arthritis | 1 | 1 | 2
Smoker [Count of Participants; unit: Participants]
  Non-Smoker | 20 | 20 | 40
  Current Cigarette Smoke | 4 | 6 | 10
  Ex Smoker | 24 | 22 | 46

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Polyethylene Inlay Wear by Roentgen Stereophotogrammetric Analysis (RSA).
Description: RSA is a highly accurate technique for the assessment of three-dimensional migration and micro motion of a joint replacement prosthesis relative to the bone it is attached to. Because of the high accuracy, RSA can also be used to measure wear in knee replacements and is used in this study for the assessment of the wear of the two polyethylene inlay types N2Vac polyethylene and X3 polyethylene.
Time Frame: 1, 2 and 5 years follow-up
Population: Negative wear values represent a decrease in liner thickness (= wear).
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | N2Vac Polyethylene Inlay | X3 Highly Cross-linked Polyethylene
Number analyzed (Participants) | 45 | 47
mm
  1 year medial wear | -0.08 (0.35) | -0.03 (0.48)
  1 year lateral wear | 0.22 (0.29) | 0.22 (0.35)
  1 year total wear | -0.03 (0.20) | -0.00 (0.26)
  2 years medial wear: number analyzed (Participants) | 45 | 45
  2 years medial wear | -0.14 (0.36) | -0.11 (0.47)
  2 years lateral wear: number analyzed (Participants) | 45 | 45
  2 years lateral wear | 0.25 (0.45) | 0.33 (0.41)
  2 years total wear: number analyzed (Participants) | 45 | 45
  2 years total wear | -0.06 (0.24) | -0.04 (0.16)
  5 years medial wear: number analyzed (Participants) | 40 | 44
  5 years medial wear | -0.23 (0.49) | -0.16 (0.47)
  5 years lateral wear: number analyzed (Participants) | 40 | 44
  5 years lateral wear | 0.14 (0.46) | 0.29 (0.47)
  5 years total wear: number analyzed (Participants) | 40 | 44
  5 years total wear | -0.23 (0.25) | -0.08 (0.17)

2. Secondary Outcome: Assessment of Prosthetic Migration Results After Two Years by RSA.
Description: RSA is a highly accurate technique for the assessment of three-dimensional migration and micro motion of a joint replacement prosthesis relative to the bone it is attached to. This study evaluates the prosthetic migration results with focus of the two years results of the Triathlon CS Peri-Apatite coated tibial and femoral components.
Time Frame: 3 and 6 months,1, 2 and 5 years follow-up
Population: The migration of the prosthesis components was calculated with a minimum of four RSA bone markers. In some cases only 3 RSA bone markers was used to calculate the migration, leading to inaccurate orientation matching of the bone markers. These patients are not included in the results describing the two different liner groups.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | N2Vac Polyethylene Inlay | X3 Highly Cross-linked Polyethylene
Number analyzed (Participants) | 46 | 47
mm
  Femur migration 3 months: number analyzed (Participants) | 42 | 45
  Femur migration 3 months | 0.723 (0.406) | 0.925 (0.516)
  Femur migration 6 months: number analyzed (Participants) | 43 | 45
  Femur migration 6 months | 0.894 (0.464) | 0.962 (0.613)
  Femur migration 1 year: number analyzed (Participants) | 42 | 45
  Femur migration 1 year | 0.912 (0.560) | 1.023 (0.741)
  Femur migration 2 years: number analyzed (Participants) | 41 | 44
  Femur migration 2 years | 0.930 (0.532) | 1.074 (0.744)
  Femur migration 5 years: number analyzed (Participants) | 35 | 42
  Femur migration 5 years | 1.078 (0.565) | 1.251 (0.810)
  Tibia migration 3 months | 0.798 (0.685) | 0.809 (0.616)
  Tibia migration 6 months | 0.873 (0.771) | 0.903 (0.677)
  Tibia migration 1 year: number analyzed (Participants) | 45 | 47
  Tibia migration 1 year | 0.975 (0.855) | 0.924 (0.662)
  Tibia migration 2 years: number analyzed (Participants) | 45 | 45
  Tibia migration 2 years | 1.043 (0.930) | 0.956 (0.681)
  Tibia migration 5 years: number analyzed (Participants) | 40 | 44
  Tibia migration 5 years | 1.039 (0.759) | 1.018 (0.673)

3. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Knee Society Score (KSS)
Description: The Knee Society Clinical Rating System is comprised of two distinct sub-scores: one for pain, range of motion (ROM) and joint stability, and one for functional parameters. Sub-scores range from a potential minimum score of 0 to a maximum score of 100 points. Although the specific scores are not distinguished as "excellent," "good," "fair," or "poor," a higher value represents a better outcome.
Time Frame: Pre-operative, 6 weeks, 3 and 6 months, 1, 2 and 5 years
Population: Participants with available data. Overall number of participants and units analyzed is based upon the preoperative population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N2Vac Polyethylene Inlay | X3 Highly Cross-linked Polyethylene
Number analyzed (Participants) | 48 | 48
units on a scale
  Pain motion score pre-operative | 49.09 (11.84) | 50.05 (15.72)
  Pain motion score 6 weeks: number analyzed (Participants) | 46 | 47
  Pain motion score 6 weeks | 68.67 (15.45) | 66.06 (15.04)
  Pain motion score 3 months: number analyzed (Participants) | 46 | 48
  Pain motion score 3 months | 77.45 (13.82) | 78.99 (15.57)
  Pain motion score 6 months: number analyzed (Participants) | 47 | 47
  Pain motion score 6 months | 82.52 (10.83) | 83.17 (13.95)
  Pain motion score 1 year: number analyzed (Participants) | 46 | 48
  Pain motion score 1 year | 84.36 (10.26) | 87.49 (9.42)
  Pain motion score 2 years: number analyzed (Participants) | 45 | 45
  Pain motion score 2 years | 82.10 (12.48) | 83.53 (14.66)
  Pain motion score 5 years: number analyzed (Participants) | 41 | 45
  Pain motion score 5 years | 82.68 (10.11) | 82.69 (9.89)
  Function score pre-op | 62.29 (15.94) | 65.10 (14.09)
  Function score 6 weeks: number analyzed (Participants) | 46 | 47
  Function score 6 weeks | 55.11 (12.53) | 51.81 (18.17)
  Function score 3 months: number analyzed (Participants) | 46 | 48
  Function score 3 months | 74.35 (12.10) | 71.67 (21.00)
  Function score 6 months: number analyzed (Participants) | 47 | 47
  Function score 6 months | 82.55 (13.44) | 82.23 (13.20)
  Function score 1 year: number analyzed (Participants) | 46 | 48
  Function score 1 year | 87.39 (14.21) | 86.98 (12.82)
  Function score 2 years: number analyzed (Participants) | 46 | 45
  Function score 2 years | 87.39 (13.54) | 83.44 (16.66)
  Function score 5 years: number analyzed (Participants) | 41 | 45
  Function score 5 years | 88.05 (12.34) | 81.33 (18.93)

4. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Short Form Patient Questionnaire (SF-36)
Description: The SF-36 Health Survey is a 36-item patient completed questionnaire to measure general health and well-being. It includes a physical and mental status component score; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: Pre-operative, 6 weeks, 3 and 6 months, 1, 2 and 5 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N2Vac Polyethylene Inlay | X3 Highly Cross-linked Polyethylene
Number analyzed (Participants) | 48 | 48
units on a scale
  Physical role functioning pre-operative: number analyzed (Participants) | 48 | 47
  Physical role functioning pre-operative | 47.40 (23.24) | 44.81 (21.20)
  Physical role functioning 6 weeks: number analyzed (Participants) | 47 | 47
  Physical role functioning 6 weeks | 30.45 (18.12) | 26.99 (18.73)
  Physical role functioning 3 months: number analyzed (Participants) | 46 | 48
  Physical role functioning 3 months | 48.91 (23.90) | 47.14 (22.64)
  Physical role functioning 6 months: number analyzed (Participants) | 47 | 48
  Physical role functioning 6 months | 61.04 (25.92) | 67.84 (22.86)
  Physical role functioning 1 year: number analyzed (Participants) | 46 | 47
  Physical role functioning 1 year | 71.06 (23.18) | 69.28 (24.89)
  Physical role functioning 2 years: number analyzed (Participants) | 46 | 46
  Physical role functioning 2 years | 68.75 (26.68) | 67.80 (24.13)
  Physical role functioning 5 years: number analyzed (Participants) | 42 | 45
  Physical role functioning 5 years | 69.49 (25.41) | 66.25 (22.77)
  Body pain pre-operative | 41.25 (16.06) | 39.33 (16.61)
  Body pain 6 weeks: number analyzed (Participants) | 47 | 47
  Body pain 6 weeks | 44.79 (21.13) | 42.40 (17.46)
  Body pain 3 months: number analyzed (Participants) | 46 | 48
  Body pain 3 months | 58.09 (20.14) | 60.13 (21.20)
  Body pain 6 months: number analyzed (Participants) | 47 | 48
  Body pain 6 months | 68.23 (21.12) | 70.15 (21.46)
  Body pain 1 year: number analyzed (Participants) | 46 | 48
  Body pain 1 year | 72.33 (22.50) | 70.65 (23.20)
  Body pain 2 years: number analyzed (Participants) | 46 | 46
  Body pain 2 years | 70.61 (23.95) | 72.93 (23.17)
  Body pain 5 years: number analyzed (Participants) | 42 | 44
  Body pain 5 years | 76.14 (24.43) | 69.14 (24.35)
  Vitality pre-operative | 60.68 (16.24) | 61.72 (18.34)
  Vitality 6 weeks: number analyzed (Participants) | 47 | 48
  Vitality 6 weeks | 59.18 (16.70) | 58.59 (16.52)
  Vitality 3 months | 68.89 (17.17) | 62.89 (17.56)
  Vitality 6 months: number analyzed (Participants) | 47 | 48
  Vitality 6 months | 70.74 (17.59) | 68.23 (17.25)
  Vitality 1 year: number analyzed (Participants) | 46 | 48
  Vitality 1 year | 71.33 (16.57) | 68.62 (19.78)
  Vitality 2 years: number analyzed (Participants) | 45 | 46
  Vitality 2 years | 71.39 (17.15) | 68.21 (18.33)
  Vitality 5 years: number analyzed (Participants) | 42 | 45
  Vitality 5 years | 70.24 (15.89) | 69.31 (18.63)
  Social role functioning pre-operative | 73.18 (22.53) | 68.23 (23.10)
  Social role functioning 6 weeks: number analyzed (Participants) | 47 | 48
  Social role functioning 6 weeks | 61.70 (23.97) | 56.25 (26.02)
  Social role functioning 3 months: number analyzed (Participants) | 46 | 48
  Social role functioning 3 months | 79.89 (21.88) | 74.22 (24.79)
  Social role functioning 6 months: number analyzed (Participants) | 47 | 48
  Social role functioning 6 months | 87.50 (17.10) | 86.20 (21.54)
  Social role functioning 1 year: number analyzed (Participants) | 46 | 48
  Social role functioning 1 year | 86.41 (18.03) | 86.46 (21.01)
  Social role functioning 2 years: number analyzed (Participants) | 45 | 46
  Social role functioning 2 years | 89.17 (17.20) | 83.15 (23.20)
  Social role functioning 5 years: number analyzed (Participants) | 42 | 44
  Social role functioning 5 years | 88.99 (17.08) | 82.10 (23.60)
  Emotional role functioning pre-operative | 78.47 (22.36) | 70.14 (29.21)
  Emotional role functioning 6 weeks: number analyzed (Participants) | 47 | 47
  Emotional role functioning 6 weeks | 67.91 (29.07) | 64.18 (34.55)
  Emotional role functioning 3 months: number analyzed (Participants) | 46 | 48
  Emotional role functioning 3 months | 75.18 (23.34) | 74.65 (29.46)
  Emotional role functioning 6 months: number analyzed (Participants) | 47 | 48
  Emotional role functioning 6 months | 80.14 (24.10) | 80.90 (23.20)
  Emotional role functioning 1 year: number analyzed (Participants) | 46 | 48
  Emotional role functioning 1 year | 84.78 (19.99) | 79.69 (26.94)
  Emotional role functioning 2 years: number analyzed (Participants) | 46 | 46
  Emotional role functioning 2 years | 84.78 (22.81) | 75.18 (27.45)
  Emotional role functioning 5 years: number analyzed (Participants) | 42 | 45
  Emotional role functioning 5 years | 85.53 (21.32) | 80.74 (22.96)
  Mental health pre-operative | 76.98 (16.79) | 75.83 (19.32)
  Mental health 6 weeks: number analyzed (Participants) | 47 | 48
  Mental health 6 weeks | 75.00 (18.96) | 76.04 (18.68)
  Mental health 3 months: number analyzed (Participants) | 46 | 48
  Mental health 3 months | 80.98 (18.61) | 77.08 (21.21)
  Mental health 6 months: number analyzed (Participants) | 47 | 48
  Mental health 6 months | 82.98 (17.74) | 81.88 (18.02)
  Mental health 1 year: number analyzed (Participants) | 46 | 48
  Mental health 1 year | 84.89 (15.41) | 78.02 (21.35)
  Mental health 2 years | 84.22 (13.78) | 77.39 (19.97)
  Mental health 5 years | 80.60 (18.23) | 80.00 (18.01)
  General health perceptions pre-op | 70.50 (17.91) | 70.44 (17.89)
  General health perceptions 6 weeks: number analyzed (Participants) | 47 | 48
  General health perceptions 6 weeks | 74.09 (15.51) | 71.13 (18.01)
  General health perceptions 3 months: number analyzed (Participants) | 46 | 48
  General health perceptions 3 months | 75.70 (17.87) | 70.56 (19.07)
  General health perceptions 6 months: number analyzed (Participants) | 47 | 48
  General health perceptions 6 months | 73.66 (17.71) | 70.23 (19.82)
  General health perceptions 1 year: number analyzed (Participants) | 46 | 48
  General health perceptions 1 year | 72.83 (16.06) | 71.92 (20.59)
  General health perceptions 2 years: number analyzed (Participants) | 46 | 46
  General health perceptions 2 years | 72.50 (16.85) | 69.63 (19.27)
  General health perceptions 5 years: number analyzed (Participants) | 42 | 45
  General health perceptions 5 years | 69.90 (16.85) | 63.76 (21.29)

5. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the EuroQuol - 5 Dimension (EQ-5D) Patient Questionnaire
Description: The EuroQol-5 Dimension (EQ-5D) is a subject-completed questionnaire designed to assess subject health state values. The EQ-5D consists of 2 areas; EQ-5D descriptive system and the visual analogue scale (VAS). The EQ-5D descriptive system comprises the following five dimensions: mobility self care, usual activities, pain/comfort and anxiety/depression. Each dimension has 3 levels indicating no problems, some problems or extreme problems. The index values on a scale between -1 (low) and 1 (high) are showing the average health status according to the 5 dimensions: A low score shows worse health and a high score shows better health.
  With the EQ VAS the respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Time Frame: Pre-operative, 6 weeks, 3 and 6 months, 1, 2 and 5 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N2Vac Polyethylene Inlay | X3 Highly Cross-linked Polyethylene
Number analyzed (Participants) | 48 | 48
units on a scale
  EQ-5D descriptive pre-operative | 0.52 (0.26) | 0.55 (0.25)
  EQ-5D descriptive 6 weeks: number analyzed (Participants) | 47 | 48
  EQ-5D descriptive 6 weeks | 0.65 (0.21) | 0.65 (0.21)
  EQ-5D descriptive 3 months: number analyzed (Participants) | 46 | 48
  EQ-5D descriptive 3 months | 0.75 (0.18) | 0.72 (0.21)
  EQ-5D descriptive 6 months: number analyzed (Participants) | 47 | 48
  EQ-5D descriptive 6 months | 0.78 (0.16) | 0.81 (0.22)
  EQ-5D descriptive 1 year: number analyzed (Participants) | 46 | 48
  EQ-5D descriptive 1 year | 0.81 (0.19) | 0.82 (0.24)
  EQ-5D descriptive 2 years: number analyzed (Participants) | 46 | 46
  EQ-5D descriptive 2 years | 0.85 (0.18) | 0.84 (0.18)
  EQ-5D descriptive 5 years: number analyzed (Participants) | 42 | 45
  EQ-5D descriptive 5 years | 0.81 (0.22) | 0.82 (0.23)
  VAS pre-operative | 68.27 (17.27) | 71.60 (14.97)
  EQ-5D VAS 6 weeks: number analyzed (Participants) | 47 | 48
  EQ-5D VAS 6 weeks | 74.49 (12.48) | 71.46 (10.45)
  EQ-5D VAS 3 months: number analyzed (Participants) | 46 | 48
  EQ-5D VAS 3 months | 76.74 (11.28) | 75.83 (11.50)
  EQ-5D VAS 6 months: number analyzed (Participants) | 47 | 48
  EQ-5D VAS 6 months | 81.26 (11.19) | 78.63 (14.65)
  EQ-5D VAS 1 year: number analyzed (Participants) | 46 | 48
  EQ-5D VAS 1 year | 81.98 (10.65) | 80.08 (14.37)
  EQ-5D VAS 2 years: number analyzed (Participants) | 46 | 44
  EQ-5D VAS 2 years | 81.76 (11.85) | 79.14 (12.38)
  EQ-5D VAS 5 years: number analyzed (Participants) | 42 | 45
  EQ-5D VAS 5 years | 79.38 (11.88) | 76.98 (12.22)

6. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With the Lower Extremity Activity Scale (LEAS) Patient Questionnaire
Description: The LEAS is completed by the participant to assess activity level. Activity levels were ordered in terms of intensity from 1 to 18, with 18 indicating the highest activity level.
Time Frame: Pre-operative, 6 weeks, 3 and 6 months, 1, 2 and 5 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | N2Vac Polyethylene Inlay | X3 Highly Cross-linked Polyethylene
Number analyzed (Participants) | 48 | 48
units on a scale
  Activity level pre-operative | 9.29 (2.69) | 8.98 (2.98)
  Activity level 6 weeks: number analyzed (Participants) | 47 | 48
  Activity level 6 weeks | 7.13 (0.64) | 7.06 (1.57)
  Activity level 3 months: number analyzed (Participants) | 46 | 48
  Activity level 3 months | 9.17 (2.39) | 8.73 (2.41)
  Activity level 6 months: number analyzed (Participants) | 47 | 48
  Activity level 6 months | 11.04 (2.67) | 11.00 (3.23)
  Activity level 1 year: number analyzed (Participants) | 46 | 48
  Activity level 1 year | 11.91 (2.41) | 11.10 (3.03)
  Activity level 2 years: number analyzed (Participants) | 46 | 46
  Activity level 2 years | 11.91 (2.98) | 11.04 (3.32)
  Activity level 5 years | 12.17 (3.34) | 10.87 (3.68)

ADVERSE EVENTS:
Time Frame: Recording of Adverse Events ongoing from when the subject has signed the informed consent up to 5 years follow-up.
Arm/Group | N2Vac Polyethylene Inlay | X3 Highly Cross-linked Polyethylene
All-Cause Mortality (participants affected / at risk) | 3/48 | 1/48
Serious Adverse Events (participants affected / at risk) | 22/48 | 24/48
Other Adverse Events (participants affected / at risk) | 3/48 | 6/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N2Vac Polyethylene Inlay (N=48) | X3 Highly Cross-linked Polyethylene (N=48)
Deep infection operatve site (Infections and infestations) | 0 (0) | 1 (1)
Delayed wound healing operative site (Surgical and medical procedures) | 1 (1) | 0 (0)
Flexion contracture operative site (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hemarthrosis after use of anticoagulant (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthrofibrosis operative site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Instability operative site (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Bradicardia (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 0 (0)
Hernia diafragmatica (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gall bladder stones (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea for 30 days (Gastrointestinal disorders) | 0 (0) | 1 (1)
Crohns Disease (Immune system disorders) | 0 (0) | 1 (1)
Collitis (Immune system disorders) | 0 (0) | 1 (1)
Infection of contralateral knee replacement (Infections and infestations) | 1 (1) | 0 (0)
Face surgery after fall accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Carpometacarpal joint 1 resection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Clavicle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ankle fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder tension rupture right (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar vertebra stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendovaginitis stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Toxic thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowel cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urothelial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Delirium (Nervous system disorders) | 1 (1) | 0 (0)
Stress incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vascular sclerosis (Vascular disorders) | 1 (1) | 1 (1)
Inguinal artery obstruction (Vascular disorders) | 0 (0) | 1 (1)
Arteria femoralis occlusion both sides (Vascular disorders) | 1 (1) | 0 (0)
Vasovagal Collapse (Vascular disorders) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N2Vac Polyethylene Inlay (N=48) | X3 Highly Cross-linked Polyethylene (N=48)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (3)
Deep vein thrombisis (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2010-07-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT02525588/Prot_SAP_000.pdf
  • Informed Consent Form (2011-09-13): https://cdn.clinicaltrials.gov/large-docs/88/NCT02525588/ICF_001.pdf